CLINICAL TRIAL: NCT03100318
Title: Benzbromarone-Controlled, Double-Blind, Comparative Study of FYU-981 for Hyperuricemia With or Without Gout to Evaluate the Safety and Noninferiority of FYU-981 (Phase III Study)
Brief Title: Benzbromarone-Controlled, Double-Blind, Comparative Study of FYU-981 in Hyperuricemia With or Without Gout
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fuji Yakuhin Co., Ltd. (Industry)
Collaborators: Mochida Pharmaceutical Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FYU-981-011
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Hyperuricemia With or Without Gout
MeSH Terms: interventions — dotinurad; Benzbromarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FYU-981 (Experimental)
  Interventions: Drug: FYU-981
- Benzbromarone (Active Comparator)
  Interventions: Drug: Benzbromarone

INTERVENTIONS:
Drug: FYU-981 — Oral daily dosing for 14 weeks
  Arms: FYU-981
Drug: Benzbromarone — Oral daily dosing for 14 weeks
  Arms: Benzbromarone

SUMMARY:
FYU-981 or Benzbromarone are administrated to hyperuricemia patients with or without gout for 14 weeks to compare the efficacy and safety of these drugs by the method of multicenter, randomized, double-blind, ascending dose regimen.

ELIGIBILITY:
Inclusion Criteria:

* Hyperuricemic or gout patients
* Serum urate level:

>= 7.0mg/dL in patients with history of gout, or >= 8.0mg/dL in patients with hypertension, diabetes or metabolic syndrome, or >= 9.0mg/dL

Exclusion Criteria:

* Gouty arthritis within two weeks before start of study treatment
* Secondary hyperuricemia
* HbA1c: >= 8.4%
* Uric acid-overproduction type in the classification of hyperuricemia
* History of, clinically significant cardiac, hematologic and hepatic disease
* Kidney calculi or clinically significant urinary calculi
* Hepatic dysfuction, or AST: >=100 IU/L or ALT: >=100 IU/L at the pre-examination
* eGFR: < 30mL/min/1.73m^2
* Systolic blood pressure: >= 180 mmHg
* Diastolic blood pressure: >= 110 mmHg

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Percent reduction from baseline in serum urate level at the final visit | 14 weeks
  Percent reduction from baseline in serum urate level at the final visit

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Tokyo, Japan

REFERENCES:
- [Derived] Hosoya T, Sano T, Sasaki T, Fushimi M, Ohashi T. Dotinurad versus benzbromarone in Japanese hyperuricemic patient with or without gout: a randomized, double-blind, parallel-group, phase 3 study. Clin Exp Nephrol. 2020 Mar;24(Suppl 1):62-70. doi: 10.1007/s10157-020-01849-0. Epub 2020 Jan 24. PMID 31980978